CLINICAL TRIAL: NCT02799238
Title: An Open Label, Randomised, Phase II Study to Investigate the Efficacy and Safety of ALECSAT Treatment as an add-on Therapy to Radiotherapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Autologuos Lymphoid Effector Cells Specific Against Tumour (ALECSAT) as Add on to Standard of Care in Patients With Glioblastoma
Acronym: ALECSAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV-006
Record Dates: First submitted 2016-06-06; First posted 2016-06-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Glioblastoma
Keywords: glioblastoma, GBM, immunotherapy, autologous lymphoid effector cells specific against tumour cells, ALECSAT, Stupp regimen, TMZ, radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy in combination with Temozolomide (TMZ) (Active Comparator): radiotherapy combined with TMZ treatment followed by adjuvant TMZ
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide
- ALECSAT + Radiotherapy in combination with TMZ (Experimental): 3 doses of ALECSAT /4 weeks followed by ALECSAT every 3 months
  Interventions: Biological: ALECSAT; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Biological: ALECSAT — 3 doses of ALECSAT/4 weeks followed by ALECSAT/3 months
  Arms: ALECSAT + Radiotherapy in combination with TMZ
Radiation: Radiotherapy — Radiotherapy 5 days/week for 6 weeks
Drug: Temozolomide — Temozolomide daily for 6 weeks followed by 6 cycles 5days/4weeks

SUMMARY:
This is a randomised, open-label, multi-centre, Phase II study in patients with newly diagnosed glioblastoma.

62 patients with newly diagnosed glioblastoma are enrolled in the study in a 1:2 allocation (standard of care (SOC): ALECSAT as an adjunct therapy to SOC).

Patients recruited into this study will receive either:

* ALECSAT as an adjunct therapy to standard of care for newly diagnosed glioblastoma (first line therapy: Stupp regimen, followed by second line therapy at the Investigator's discretion) or
* Standard of care therapy for newly diagnosed glioblastoma (first line therapy: Stupp regimen, followed by second line therapy at the Investigator's discretion).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged between 18 and 70.
* Histologically confirmed glioblastoma (Grade IV) diagnosis.
* Eligible for combined radiotherapy and TMZ treatment.
* Patients with complete or partial tumour resection. For patients with limited tumour volume, biopsy is acceptable.
* WHO Performance status 0-2.
* Body weight ≥ 40 kg (males), ≥ 50 kg (females).
* Able and willing to provide written informed consent and comply with the study protocol and procedures.
* Women of child-bearing potential must have a negative pregnancy test at screening and agree to use acceptable methods of contraception during the trial.

Exclusion Criteria:

* Prior treatment for brain tumours at study entry.
* Prior treatment with temozolomide at study entry.
* Females who are pregnant, planning to become pregnant or breastfeeding.
* Positive tests for anti- human immunodeficiency virus (HIV)-1/2; HBsAg, anti HBc, anti-HCV or being positive in a Treponema Pallidum test (syphilis).
* Patients who may have been exposed to West Nile virus or Dengue fever virus within the last 28 days prior to enrolment or Ebola virus within the last 60 days prior to enrolment should be excluded, unless the patient has been tested negative.
* Patients from high incidence areas for Human T-Lymphotropic Virus (HTLV-1) virus or who has a parent or spouse from a high incidence area must be excluded unless tested negative for HTLV-1 virus.
* Known allergy to study medication.
* Any condition or illness that, in the opinion of the Investigator or medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the investigational drug.
* Any concurrent illness that may worsen or cause complications in connection with blood donation, for example uncontrolled epilepsy, cardiovascular, cerebrovascular or respiratory disease.
* Use of immunosuppressant drugs with the exception of steroids. Blood transfusion within 48 hours prior to the donation of blood for ALECSAT production.
* Low haemoglobin count in the opinion of the Investigator.
* Lymphocyte count <0.3 x 109/litre.
* Participation in any other interventional clinical trial within 30 days prior to inclusion.
* TMZ contraindication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months after LPFV or when 47 patients has reached investigator assessed disease progression or death from any cause
  Compare the progression free survival between patients who receive ALECSAT as add on to SoC and patients who only receive SoC

SECONDARY OUTCOMES:
Proportion of patients alive at 12 and 24 months | 24 months after LPFV or when 47 patients has reached investigator assessed disease progression or death from any cause
  To compare OS rate at 12 and 24 months between patients who receive ALECSAT as add on to SoC and patients who only receive SoC
Frequency and Severity of treatment related Adverse Events | Up to 24 months after randomisation of last patient
  Comparison of frequency and severity of treatment related AEs in the 2 study groups

CONTACTS AND LOCATIONS:
Overall Officials: Katja Werlenius, PhD, Principal Investigator — Sahlgrenska University Hospital, Gothenburg
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Ryhov hospital, Jönköping
  - Skånes university hospital, Lund
  - Karolinska University hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No